CLINICAL TRIAL: NCT07260383
Title: Enhancing Home-Based Exercise Therapy With Telerehabilitation in Mild Adolescent Idiopathic Scoliosis: A Randomized Controlled Trial
Brief Title: Telerehabilitation Support for Home Exercise in Mild AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZDT--2025
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis Idiopathic; Telerehabilitation; Exercise
Keywords: scoliosis; telerehabilitation; Home-based exercise
MeSH Terms: conditions — Motor Activity; Scoliosis | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Exercise (Active Comparator)
  Interventions: Procedure: home exercise
- Telerehabilitation (Active Comparator)
  Interventions: Procedure: telerehabilitation

INTERVENTIONS:
Procedure: home exercise — Self Scoliosis exercises. home exercises were shown to the control group and a form containing explanations and pictures of the exercises was shared with the patient in printed form. They are very common well known posture exercises including postural correction, strengthening and core stabilization. Participants were asked to apply the exercises at least three times a week and to record the day and duration of each exercise session in. an exercise diary. The researcher physiotherapist called these participants every two weeks to follow their compliance with the exercise program. At the end of the eight-week application period, the participants were invited back to the clinic and re-evaluated with the same evaluation methods.
  Arms: Home-based Exercise
Procedure: telerehabilitation — Patient specific exercises with supervised telerehabilitation. Participants included in the study program group also had the same home exercise program given in the hospital. The exercises were same with the other group. In addition to these home exercises, the exercises were done online under the guidance of a physiotherapist once a week. An appointment was made for the first telerehabilitation session for the patients in the study group after the evaluation and the same exercise form was shared with this group. In the online sessions, whether the patient correctly applied the exercise program defined for him/her was monitored and checked online once a week
  Arms: Telerehabilitation

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional spinal deformity that affects postural alignment, function, and quality of life. Telerehabilitation has emerged as a promising approach to enhance accessibility and continuity of exercise-based treatment in AIS. This study aimed to compare the effects of telerehabilitation-supported home exercise programs with standard home exercises on posture, pain, body image, and quality of life in adolescents with mild AIS.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional deformity character-ized by a curvature of the spine greater than 10 degrees in the coronal plane, a deteri-oration in the physiological curvature in the sagittal plane and accompanying rotation in the axial plane. AIS is mostly seen at the thoracic level, less frequently at the lumbar and thoracolumbar levels, and is the most common form of structural scoliosis, accounting for approximately 80% of all scoliosis cases .

In AIS, the problem with spinal alignment affects the bones and soft tissue in the entire body; the resulting deformities such as postural disorders and loss of flexibility of the spine cause problems such as cosmetic concerns, functional losses, and pain in adolescents. In severe cases, respiratory functions and lung capacity decrease, and the patient's quality of life is affected by this condition. Different treatment approaches are recommended for the prevention and management of all these problems. When determining the appro-priate treatment option, the type, shape, degree of the curve, and the patient's charac-teristics should be taken into consideration. To stop or prevent the progression of the curve or to combat the complications experienced; different exercise approaches for scoliosis, the use of corsets, and, in more severe cases, surgical methods are the basic/ main treatment options. In addition, the incidence of curves of 10° and above varies between 1 and 3%, and most of them do not require surgical intervention. For moderate curves below 40°, special exercises and corsets are expressed as first-line treatments to control scoliosis without the need for surgery, therefore various exercise approaches are frequently used at all stages of AIS treatment.

When the literature is examined, it has been reported that exercises for AIS are often recommended to prevent the progression of the curve, correct postural behavior and provide awareness, increase neuromotor control of the spine, increase spinal and thoracic flexibility, increase muscle strength by optimizing muscle balance, and achieve body symmetry. In the treatment of scoliosis, specific exercises are usually given to the individual according to the shape, type, and degree of the curve. Therapeutic exercises include breathing exercises, self-correction exercises (mental imagery, exteroceptive, proprioceptive stimuli, and mirror control), and stabilization exercises (physical exercise, yoga, pilates, and core stabilization).

Telerehabilitation-based interventions are preferred to continue treatment when patients' access to rehabilitation needs is restricted for various reasons. Telerehabilitation has been applied to various diseases and has achieved significant success these days, but telerehabilitation studies in AIS patients are quite rare. Studies in this field have increased their popularity with the rise of telerehabilitation after the pandemic period and have begun to show promising results.

There are limited studies comparing telerehabilitation with home exercises; however, recent studies have shown that telerehabilitation may provide more positive results in terms of respiratory function, flexibility and participation . These findings reveal that telerehabilitation may positively affect exercise compliance and clinical out-comes in AIS; however, due to the small number of studies and the variety of exercises applied in the studies, the number of comparative data regarding the application of ex-ercises for scoliosis via telerehabilitation remains quite limited. In addition, the difference between the results obtained when the home programs are completely applied by oneself and the results obtained when a physiotherapist guides them remotely via telerehabil-itation has not been fully established. In this context, the aim of the study is to examine the effectiveness of the home-based exercise program, which is recommended as a standard after diagnosis in the hospital, in individuals diagnosed with adolescent idiopathic sco-liosis (AIS) and supported by a physiotherapist via telerehabilitation, compared to the same exercise program being applied individually at home. Our study is one of the few that directly examines the effect of supervision on clinical outcomes and has a unique place in terms of comparative evaluation of telerehabilitation with home programs.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study were "being between 10 and 18 years old, di-agnosed with adolescent idiopathic scoliosis (AIS) and not using a corset, having a Risser stage between 0 and 3 and a Cobb angle between 10° and 25°, individuals with a Type I curve pattern according to the Lenke classification."

Exclusion Criteria:

The exclusion criteria were determined as "those with any medical contraindication that may prevent them from doing exercise, patients who have undergone any treatment for scoliosis within the last year, patients who have undergone spinal surgery and patients using a corset, and patients with any mental, neurological and pulmonary disease."

-

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2025-09-13 (Actual)

PRIMARY OUTCOMES:
Newyork posture scale | baseline and week 8
Walter Reed Visual Assessment Scale | Baseline and week 8
cobb angle | baseline
visual analog scale | baseline and week 8
Scoliosis Research Society -22 (srs 22) | baseline and week 8

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No